CLINICAL TRIAL: NCT05275959
Title: Implementation Research on the Construction and Scale Up Regarding To"Comorbidity-Co-causes-Joint-prevention" Comprehensive Demonstration District of Myopia and Obesity Among Children and Adolescents in Beijing Guided by RE-AIM Framework
Brief Title: Beijing (Peking)---Myopia and Obesity Comorbidity Intervention (BMOCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Yi Song2022
Record Dates: First submitted 2022-01-20; First posted 2022-03-11 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Myopia
Keywords: Children; Adolescents; Myopia; Obesity; Cluster randomized controlled trial
MeSH Terms: conditions — Obesity; Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "22510SS" Intervention (Other): Intervention measures will be taken against children and adolescents' myopia and obesity at four levels: individual (individual centered activities), environment (supportive family and school settings), and supervision (family, school, program team, and clinical) and feedback (timely feedback from the WeChat applet).
  Interventions: Other: A cluster randomized trial of a comprehensive intervention nesting family and clinic into school centered implementation to reduce myopia and obesity among children and adolescents in Beijing, China
- Control (No Intervention): Regular health education without extra intervention

INTERVENTIONS:
Other: A cluster randomized trial of a comprehensive intervention nesting family and clinic into school centered implementation to reduce myopia and obesity among children and adolescents in Beijing, China — Myopia and obesity in children and adolescents have become serious public health problems that endanger public health, especially in China. Unhealthy lifestyle behaviors are environmental drivers of both myopia and obesity. This protocol describes a study to evaluate the effectiveness of "22510SS", that is 2 h of daytime outdoor activities ('2'); Limit screen time to no more than 2 h per day ('2'); Consume at least 5 servings of fruits and vegetables daily ('5'); Attain 1 h of physical activity daily ('1'); Consume 0 sugar-sweetened beverages ('0'); Reasonable sleep duration ('S'); Regular supervision ('S'). A school-based, multifaceted intervention strategy for myopia and obesity prevention, and to assess and explore the implementation of "22510SS" with regards to acceptability, feasibility, adoption, usage and maintenance.
  Other Names: Myopia and Obesity Comorbidity intervention
  Arms: "22510SS" Intervention

SUMMARY:
Based on the RE-AIM framework, this project intends to integrate the prevention and control measures of myopia and obesity, and establish a set of key suitable technical packages and guarantee systems for the "comorbidity-common-cause-common prevention" of myopia and obesity in children and adolescents. Dong cheng ,Tongzhou and Changping District in total selected 18 intervention schools and 18 control schools to apply the application, integrate the resources of the "family-school-community-medical institution", and establish a comprehensive combination of myopia and obesity in children and adolescents In the prevention and control demonstration area, intervention study was conducted to evaluate the comprehensive intervention effect of myopia and obesity in children and adolescents in the demonstration area, and to promote it through the regional monitoring system in Beijing. This project is the first time to establish a district-level comprehensive prevention and control demonstration area for children and adolescents with myopia and obesity that can be promoted, including key appropriate technology packages and promotion and application strategies. Healthy Beijing 2030" plan laid the foundation.

DETAILED DESCRIPTION:
Baseline (March-April 2023), first follow-up (July-August 2023), and second follow-up (November-December 2023). The collection of data from study participants at baseline and third follow-up included questionnaire collection, anthropometric indicators, body composition measurements, vision measurements, blood pressure measurements, urine, saliva, and venous blood draws, as well as home questionnaires, school questionnaires, and interventionist physician questionnaires from the community hospitals and the project hospitals; and the first follow-up (the collection of data varied in each district, and was done according to the level of district cooperation) included questionnaire collection, anthropometric measurements, vision measurements, and blood pressure measurements, as well as home questionnaires, school questionnaires, and interventionist physician questionnaires from the community hospitals and the project hospitals.

Myopia and activity records: including nighttime lighting, wake-sleep cycles, and movement. As well as family questionnaires, school questionnaires, community hospitals and project hospital intervention doctor questionnaires. All inspection items are operated by trained and qualified doctors and professional health technicians. The inspection will be arranged in the school, and the whole process is the same as the regular physical examination in the school.

The child required 2 venous blood collections, urine and saliva collections during the year (at the initial stage and at the 3rd follow-up, respectively).

Blood sample testing: 10ml of venous blood is drawn each time for blood routine and blood biochemistry. The blood process is safe. Blood samples include: blood biochemical indicators (fasting blood glucose (FBG), insulin, total cholesterol (TC), triglyceride (TG), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C) ) and so on).

Hormone testing: Collect saliva samples in the morning and purchase ELISA kits to measure levels of thyroid hormones, estradiol and testosterone.

Urine sample testing: use polypropylene urine cups and urine collection tubes (without PAEs plasticizers) to collect 10 mL of urine from the research subjects, and reserve the sample to collect the first excretion after getting up in the morning, before breakfast and before exercising. The collected urine samples were uniformly stored in a 5mL centrifuge tube and stored in a -20°C refrigerator. Urine PAEs and their metabolites: Ultra-high performance liquid chromatography-tandem mass spectrometry (UPLC-MS/MS) was used to detect seven PAEs metabolites in students' urine: monomethyl phthalate (MMP), phthalic acid Monoethyl ester (MEP), mono-n-butyl phthalate (MBP), mono(2-ethylhexyl) phthalate (MEHP), mono(2-ethyl-5-phthalate) Hydroxyhexyl) ester (MEHHP), mono(2-ethyl-5-oxohexyl) phthalate (MEOHP).

The content of the family and student questionnaires will include general conditions of children, general conditions of parents and families, as well as daily diet, physical activity and sleep. The name of the child will only be used for tracking and will be deleted after one year of observation to ensure that the information of the child and participants will not be leaked. All members of the project team have signed a confidentiality agreement, and all information in the questionnaire will not be leaked to the outside world.

ELIGIBILITY:
Inclusion Criteria:

1. At 6-14 years old。
2. The physical examination information at school is complete.
3. There is no transfer plan within one year.

Exclusion Criteria:

1. There are ophthalmic device diseases, such as keratitis, corneal ulcer, etc.;
2. History of ophthalmic surgery, such as laser surgery;
3. Visual problems such as color weakness and color blindness;
4. History of heart disease, hypertension, diabetes, tuberculosis, asthma, hepatitis, or nephritis;
5. Obesity caused by endocrine diseases or side effects of drugs;
6. Abnormal physical development, such as dwarfism or gigantism;
7. Can not participate in school sports activities;
8. Have any weight loss behaviors such as inducing vomiting or taking weight loss drugs in past three months;
9. Body deformities, such as severe scoliosis, chicken breasts, limps, pronounced O-or X-legs.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3963 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Myopia changes | Approximate timing: Approximate timing: Measured in the baseline and the twelfth month of intervention
  Refer to the "Guidelines for the Prevention and Control of Myopia in Children and Adolescents" issued by the National Health Commission in 2019 to check the vision of children. Unaided distance visual acuity should be measured from a standard distance (5 m), using a standard chart of Illiterate E with a white background. The reduced VA was defined as the measurement value of less than 5.0 in either eye. Then, myopia was defined when participants had reduced VA and had spherical equivalent (SE) less than -0.50 D using non-cycloplegic and subjective refraction. Mild myopia was defined as the SE less than -0.50 D but greater than or equal to -3.00 D, moderate myopia was defined as less than -3.00 D but greater than or equal to -6.00 D, and severe myopia was defined as less than -6.00 D.
Height changes | Approximate timing: Approximate timing: Measured in the baseline and the twelfth month of intervention
  The record is in centimeters and accurate to one decimal place.
Weight changes | Approximate timing: Approximate timing: Measured in the baseline and the twelfth month of intervention
  Use an electronic scale and check its accuracy and sensitivity before use. The accuracy error shall not exceed 0.1%, that is, the error per 100kg shall be less than 0.1kg.
Waist circumference changes | Approximate timing: Approximate timing: Measured in the baseline and the twelfth month of intervention
  A tape ruler was used to measure horizontally around the midpoint of the line between the anterior superior iliac crest and the lower edge of the 12th rib (the thickest part of the waist was selected for obese patients);
Hip circumference changes | Approximate timing: Approximate timing: Measured in the baseline and the twelfth month of intervention
  The subject stands naturally, with the arms drooping and moderately spread, the feet together, the legs are evenly weighted, the hips are relaxed, and the eyes are straight ahead. The tester places the tape on the most protruding part of the back of the buttocks, and circles the buttocks horizontally. During the test, the tape measure should be close to the skin, and the soft tissue should not be pressed. The reading should be taken when the subject exhales calmly. To ensure that the position of the tape ruler is correct, you can move the tape ruler up and down, compare the readings at different positions, and record the maximum value.
Body composition changes | Approximate timing: Approximate timing: Measured in the baseline and the twelfth month of intervention
  The body composition measurement was conducted using the Tanita BC-420 body composition analyzer, which collects data on body fat percentage. The participants stood on the foot electrodes of the analyzer and held the hand electrode firmly while maintaining a stable posture throughout the process. The measurement was completed using the bio-electrical impedance method, which typically took between 40 to 60 seconds to obtain accurate readings of the aforementioned body composition metrics.
Blood pressure changes | Approximate timing: Approximate timing: Measured in the baseline and the twelfth month of intervention
  The upper arm medical electronic sphygmomanometer is used to measure blood pressure. During the measurement, the cuff of the sphygmomanometer is securely wrapped around the upper arm at the level of the heart, ensuring a proper fit without constriction. The device is then activated to inflate the cuff, applying pressure to the brachial artery until the pulse is no longer detectable. The pressure is gradually released, and the device records the systolic pressure (the maximum pressure in the arteries during the heart's contraction) and the diastolic pressure (the minimum pressure in the arteries during the heart's relaxation).
Blood glucose change | Approximate timing: Measured in the baseline and the twelfth month of intervention
  Blood glucose analysis was conducted using a professional method to evaluate the blood sample. First, a skilled nurse performed venipuncture to collect the blood samples from the participants. The collected blood samples were immediately frozen and stored in a -80℃ freezer until all samples were gathered for unified delivery to the laboratory. The blood samples were sent to a specialized testing center for analysis and result feedback.
Total cholesterol change | Approximate timing: Measured in the baseline and the twelfth month of intervention
  Total cholesterol analysis was conducted using a professional method to evaluate the blood sample. First, a skilled nurse performed venipuncture to collect the blood samples from the participants. The collected blood samples were immediately frozen and stored in a -80℃ freezer until all samples were gathered for unified delivery to the laboratory. The blood samples were sent to a specialized testing center for analysis and result feedback.
Low-density lipoprotein cholesterol (LDL-C) change | Approximate timing: Measured in the baseline and the twelfth month of intervention
  Low-density lipoprotein cholesterol (LDL-C) was conducted using a professional method to evaluate the blood sample. First, a skilled nurse performed venipuncture to collect the blood samples from the participants. The collected blood samples were immediately frozen and stored in a -80℃ freezer until all samples were gathered for unified delivery to the laboratory. The blood samples were sent to a specialized testing center for analysis and result feedback.
High density lipoprotein cholesterol (HDL-C) change | Approximate timing: Measured in the baseline and the twelfth month of intervention
  High density lipoprotein cholesterol (HDL-C) change was conducted using a professional method to evaluate the blood sample. First, a skilled nurse performed venipuncture to collect the blood samples from the participants. The collected blood samples were immediately frozen and stored in a -80℃ freezer until all samples were gathered for unified delivery to the laboratory. The blood samples were sent to a specialized testing center for analysis and result feedback.
Triglycerides change | Approximate timing: Measured in the baseline and the twelfth month of intervention
  Triglycerides was conducted using a professional method to evaluate the blood sample. First, a skilled nurse performed venipuncture to collect the blood samples from the participants. The collected blood samples were immediately frozen and stored in a -80℃ freezer until all samples were gathered for unified delivery to the laboratory. The blood samples were sent to a specialized testing center for analysis and result feedback.
Uric acid change | Approximate timing: Measured in the baseline and the twelfth month of intervention
  Uric acid was conducted using a professional method to evaluate the blood sample. First, a skilled nurse performed venipuncture to collect the blood samples from the participants. The collected blood samples were immediately frozen and stored in a -80℃ freezer until all samples were gathered for unified delivery to the laboratory. The blood samples were sent to a specialized testing center for analysis and result feedback.
Saliva test | Approximate timing: Approximate timing: Measured in the baseline and the twelfth month of intervention
  Professional salivary hormone detection methods were employed to analyze the saliva samples from participants. First, participants were instructed to collect saliva samples at a specified time point, typically upon waking in the morning. Collected saliva samples were stored in sterile containers and refrigerated promptly to prevent hormone degradation. Estradiol was measured from the saliva sample. The testing methods utilized high-sensitivity enzyme-linked immunosorbent assays (ELISA) to ensure precise and reliable results.
Urine sample detection changes | Approximate timing: Approximate timing: Measured in the baseline and the twelfth month of intervention
  Use polypropylene urine cups and urine collection tubes (without PAEs plasticizers) to collect 10 mL of urine from the research subjects, and reserve the sample to collect the first excretion after getting up in the morning, before breakfast and before exercising. The collected urine samples were uniformly stored in a 5mL centrifuge tube and stored in a -20°C refrigerator. Urine PAEs and their metabolites: Ultra-high performance liquid chromatography-tandem mass spectrometry (UPLC-MS/MS) was used to detect seven PAEs metabolites in students' urine: monomethyl phthalate (MMP), phthalic acid Monoethyl ester (MEP), mono-n-butyl phthalate (MBP), mono(2-ethylhexyl) phthalate (MEHP), mono(2-ethyl-5-phthalate) Hydroxyhexyl) ester (MEHHP), mono(2-ethyl-5-oxohexyl) phthalate (MEOHP).
Sleep diary | Approximate timing: Measured in the six month of intervention
  To understand students' sleep duration, data collection was conducted using sleep diaries. Each participant was required to record at least one school day and one weekend day consecutively. The sleep diary primarily recorded bedtime, actual sleep onset time, and morning wake-up time. These data were used to calculate total sleep duration per night.
Night lighting changes | Approximate timing: Measured in the third month of intervention
  Put the photometer on the bedside table of the bedroom and program it to continuously collect light information every 60 seconds.
Basic information-for student | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of student questionnaire, which was filled by students or with the help of their parents. Basic information includes students' school, grade, class, name, gender, and date of birth.
Knowledge mastery-for student | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of student questionnaire, which was filled by students or with the help of their parents. The knowledge mastery part assessing health knowledge focus on whether students can distinguish behaviors include key message of '22510ss' that promote health. Responses were categorized as "Correct" "Incorrect" or "Don't Know" The total score is the sum of each item (0 to 7), "Correct" for 1 point, and "Incorrect" "Don't Know" for 0 point. A higher total score indicates a better understanding of health knowledge.
Behavior practice-for student | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of student questionnaire, which was filled by students or with the help of their parents. The health behavior section of the questionnaire surveys students on their screen time, consumption of fruits and vegetables, intake of high-quality protein, frequency of consuming sugary drinks, and frequency of vision and weight measurement. We calculate the score of '22510ss' key healthy behavior based on their questionnaire results. Each behavior earns one point for completion, and the total score for the items is calculated. The highest score is 7 points, and the lowest is 0 point. Higher points indicate stronger health action capabilities among students.
Myopia and obesity intervention promotion/barrier factors-for student | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of student questionnaire, which was filled by students or with the help of their parents. This section of the questionnaire investigates factors that promote or hinder students' implementation of healthy behaviors, including school support, family influence, and peer influence. A five-point Likert scale ("Strongly Agree" is scored 5 points, and "Strongly Disagree" is scored 1 point) is used, and if more than 75% of respondents choose "Agree" or "Strongly Agree," the factor is considered to have a strong promoting or hindering effect.
Dietary questionnaire-for student | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of student questionnaire, which was filled by students or with the help of their parents. We used DQQ-China (Dietary Quality Questionnaire for China) to assess the dietary quality of student. DOQ collects dietary consumption data from 29 food groups and is used to calculate the Global Dietary Recommendation (GDR) score. The GDR score ranges from 0 to 18 and reflects adherence to the global dietary guidelines proposed by the World Health Organization (WHO). Higher GDR scores indicate better adherence to WHO's global dietary recommendations. Dietary quality classification based on the GDR score is as follows: High dietary quality: GDR ≥ 10; Moderate dietary quality: 8 ≤ GDR < 10; Low dietary quality: GDR < 8.
Physical activity questionnaire-for student | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of student questionnaire, which was filled by students or with the help of their parents. International Physical Activity Questionnaire (IPAQ) was used to assess physical activity levels, which includes the frequency, duration, and intensity of physical activities such as walking, moderate-intensity activities, and vigorous-intensity activities over the past 7 days, and the long form providing a more detailed assessment over a longer period. The total physical activity score was usually calculated in terms of MET-minutes/week (Metabolic Equivalent of Task), Based on the MET values (<600, 600-1500, >1500), students' activity levels are classified as low, moderate, or high.
Sleep questionnaire-for student | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of student questionnaire, which was filled by students or with the help of their parents. The Center for Epidemiologic Studies Depression Scale (CES-D) was employed, each question on the MEQ-5 is answered on a scale that reflects the degree of preference for morning or evening activity. The scores from the five items are summed up to generate an overall score that reflects the individual's chronotype: The total score of the MEO-5 ranges from 4 to 25. The scoring categories are as follows: 4-7 points: Definitely Evening Type; 8-11 points: Moderately Evening Type; 12-17 points: Intermediate Type; 18-21 points: Moderately Morning Type;22-25 points: Definitely Morning Type.
Mental health questionnaire-for student | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of student questionnaire, which was filled by students or with the help of their parents. The Center for Epidemiologic Studies Depression Scale (CES-D) was employed to assess the frequency and severity of depressive symptoms The CES-D consists of 20 items using a 4-point Likert scale (0 = "Rarely or none of the time," 3 = "Most or all of the time"). Scores for each item are summed, with higher total scores indicating more severe depressive symptoms. The total score ranges from 0 to 60. Generally, a score of 16 or higher is considered indicative of clinically significant depressive symptoms.
Basic information -for patents | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of parents' questionnaire. Basic information includes their child's school, grade, class, name, gender, and date of birth, as well as their relationship, sibling information, birth information of the child, and the parents' age.
Myopia and obesity status-for patents | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of parents' questionnaire. This section surveys the height, weight, vision status, and the presence of diseases such as hypertension and diabetes in the father and mother.
Knowledge mastery-for patents | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of parents' questionnaire. The knowledge mastery part assessing health knowledge focus on whether students can distinguish behaviors include key message of '22510ss' that promote health. Responses were categorized as "Correct" "Incorrect" or "Don't Know" The total score is the sum of each item (0 to 7), "Correct" for 1 point, and "Incorrect" "Don't Know" for 0 point. A higher total score indicates a better understanding of health knowledge.
Behavior practice-for patents | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of parents' questionnaire. The health behavior section of the questionnaire surveys parents on their screen time, consumption of fruits and vegetables, intake of high-quality protein, frequency of consuming sugary drinks, and frequency of vision and weight measurement. We calculate the score of '22510ss' key healthy behavior based on their questionnaire results. Each behavior earns one point for completion, and the total score for the items is calculated. The highest score is 7 points, and the lowest is 0 point. Higher points indicate stronger health action capabilities among students.
Child sleep quality-for patents | Approximate timing: Measured in the baseline and the twelfth month of intervention
  This is part of parents' questionnaire. This section of the questionnaire surveys parents about their child's sleep performance using Sleep Disturbance Scale for Children (SDSC). The SDSC consists of 26 items that cover various aspects of sleep, categorized into different domains, it uses a 5-point Likert scale (1 = "never," 5 = "always"), where parents report how often their child experiences each symptom. The scores are summed to generate a total score and sub-scores for each domain. Total score range of 26 to 130, we used the following thresholds to classify the severity of sleep disturbances: Score < 38: Considered no significant sleep disturbance; Scores between 38 and 45: Mild sleep disturbance; Score > 45: Significant sleep disturbance.
Basic information -for doctors of school | Approximate timing: Measured in the sixth month of intervention
  This is part of school questionnaire. Basic information includes the school doctors' gender, age, education level, and workplace.
Promotion/barrier factors in health working --for doctors of school | Approximate timing: Measured in the sixth month of intervention
  This is part of school questionnaire. We investigated the promoting and hindering factors in schools' efforts to improve students' health behaviors, including items such as the school's educational philosophy, school environment, and level of school support. The items are scored using a 5-point Likert scale ("Strongly Agree" is scored 5 points, and "Strongly Disagree" is scored 1 point). If more than 50% of school doctors select "Strongly Agree" for a particular item, it is considered an important promoting or hindering factor.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Tongzhou District Primary and Secondary School Health Care Institute, Beijing, Beijing Municipality
  - Dongcheng Primary and Secondary School Health Care Center, Beijing
  - Health Education Center forPrimary and Secondary Schools Changping, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Dang J, Liu J, Liu Y, Wang Y, Shi D, Chen Z, Yuan W, Cai S, Mi J, Xiao P, Li L, Fan Y, Gao A, Chen H, Zhuang L, Yu Z, Li J, Yang D, Yang G, Guo L, Li Y, Song J, Li J, Ma J, Dong Y, Song Y. A cluster randomized trial of a comprehensive intervention nesting family and clinic into school centered implementation to reduce myopia and obesity among children and adolescents in Beijing, China: study protocol. BMC Public Health. 2023 Jul 27;23(1):1435. doi: 10.1186/s12889-023-16270-x. PMID 37501063